

Cymru **University Hospital** 



IRAS ID: 238464 Study ID Number:

Participant Identification Number:

## **CONSULTEE DECLARATION FORM** [Version 2.0 30/01/18]

| Title of Project: Measuring Ph | ysical Activity Levels | in Critical Care: A Feasibility Stu | udy |
|---|---|---|---|
| Name of Researcher: Mrs Laur | a Jones, Dr Harriet S | hannon<br>Please initial t | юх |
| participation in this research project | | e read and understand the | |
| information sheet dated 30/01/201 the opportunity to consider the info answered satisfactorily. | | | |
| 2. In my opinion he/she would hav | e no objection to takir | ng part in the above study. | |
| 3. I understand that I can request I without giving any reason and with | | | |
| 4. I understand that relevant section during the study may be looked at UHB, University College London a | by responsible individ | duals from Cardiff and Vale | |
| relevant to their taking part in this | | | |
| 5. I agree for any data already coll study | ected to be used for t | he purposes of this research | |
| Name of Consultee | Date | Signature | _ |
| Relationship to participant: | | | |
| Person undertaking consultation (if different from researcher) | Date | Signature | _ |
| Researcher | <br>Date | <br>Signature | |

When completed: 1 (original) to be kept in medical notes, 1 for consultee; 1 for researcher site file